CLINICAL TRIAL: NCT02877927
Title: A Phase 3 Randomized, Double-Blind, Multi-Center Study to Compare the Safety and Efficacy of Oral Omadacycline to Oral Linezolid for Treating Adult Subjects With Acute Bacterial Skin and Skin Structure Infection (ABSSSI)
Brief Title: Oral Omadacycline vs. Oral Linezolid for the Treatment of ABSSSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTK0796-ABSI-16301
Record Dates: First submitted 2016-08-15; First posted 2016-08-24 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Bacterial Infections; Skin Structures and Soft Tissue Infections
MeSH Terms: conditions — Bacterial Infections; Soft Tissue Infections | interventions — omadacycline; Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omadacycline (Experimental): Omadacycline tablets
  Interventions: Drug: Omadacycline
- Linezolid (Active Comparator): Linezolid tablets
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Omadacycline — po tablets
  Arms: Omadacycline
Drug: Linezolid — po tablets
  Other Names: Zyvox
  Arms: Linezolid

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of omadacycline as compared to linezolid in the treatment of adults with acute bacterial skin and skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients, ages 18 years or older who have signed the informed consent
* Has a qualifying skin and skin structure infection
* Female patients must not be pregnant at the time of enrollment
* Must agree to a reliable method of birth control during the study and for 30 days following the last dose of study drug

Exclusion Criteria:

* Infections where the outcome is strongly influenced by factors other than protocol-defined treatments and procedures, or that require antibacterial treatment for greater than 14 days
* Evidence of significant immunological disease
* Severe renal disease or requirement for dialysis
* Evidence of septic shock
* Has a history of hypersensitivity or allergic reaction to any tetracycline or to linezolid
* Has received an investigational drug within the past 30 days
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 735 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05-26 (Actual); Study Completion 2017-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Manley, Study Director — Senior Director, Clinical Operations
Locations (50):
- United States (50):
  - Site 620, Birmingham, Alabama
  - Site 642, Mobile, Alabama
  - Site 616, Anaheim, California
  - Site 601, Anaheim, California
  - Site 636, Bakersfield, California
  - Site 606, Buena Park, California
  - Site 604, Chula Vista, California
  - Site 659, Huntington Beach, California
  - Site 608, La Mesa, California
  - Site 618, Laguna Hills, California
  - Site 612, Long Beach, California
  - Site 648, Modesto, California
  - Site 610, Oceanside, California
  - Site 615, San Diego, California
  - Site 621, San Diego, California
  - Site 613, San Francisco, California
  - Site 603, Stockton, California
  - Site 650, Torrance, California
  - Site 646, Ventura, California
  - Site 614, DeLand, Florida
  - Site 655, Fort Myers, Florida
  - Site 656, Homestead, Florida
  - Site 631, Miami, Florida
  - Site 658, Miami, Florida
  - Site 654, Miami, Florida
  - Site 626, Miami, Florida
  - Site 637, Miami, Florida
  - Site 653, Miami, Florida
  - Site 641, Miami, Florida
  - Site 645, Miami, Florida
  - Site 640, Miami Lakes, Florida
  - Site 662, Miami Lakes, Florida
  - Site 609, Saint Cloud, Florida
  - Site 644, Council Bluffs, Iowa
  - Site 657, Boston, Massachusetts
  - Site 617, St Louis, Missouri
  - Site 602, Butte, Montana
  - Site 623, Las Vegas, Nevada
  - Site 630, Somers Point, New Jersey
  - Site 647, Jackson Heights, New York
  - Site 632, Mount Airy, North Carolina
  - Site 649, Toledo, Ohio
  - Site 607, Rapid City, South Dakota
  - Site 635, Jackson, Tennessee
  - Site 628, Smyrna, Tennessee
  - Site 633, Baytown, Texas
  - Site 605, Channelview, Texas
  - Site 625, Houston, Texas
  - Site 627, Houston, Texas
  - Site 634, Sugar Land, Texas

REFERENCES:
- [Derived] Rodriguez GD, Warren N, Yashayev R, Chitra S, Amodio-Groton M, Wright K. Intravenous Versus Oral Omadacycline or Linezolid for Acute Bacterial Skin and Skin Infections: A post hoc Analysis of the OASIS Trials. Infect Dis Ther. 2024 Dec;13(12):2637-2648. doi: 10.1007/s40121-024-01057-3. Epub 2024 Oct 26. PMID 39461915
- [Derived] Vacalis S, Brunton S, Gindi J. Omadacycline in Skin Infections and Pneumonia: A Review of the Evidence. J Fam Pract. 2022 Jun;71(5 Suppl):S10-S21. doi: 10.12788/jfp.0424. PMID 35776862
- [Derived] Pai MP, Wilcox MH, Chitra S, McGovern PC. Safety and efficacy of omadacycline by BMI categories and diabetes history in two Phase III randomized studies of patients with acute bacterial skin and skin structure infections. J Antimicrob Chemother. 2021 Apr 13;76(5):1315-1322. doi: 10.1093/jac/dkaa558. PMID 33458763
- [Derived] Cornely OA, File TM Jr, Garrity-Ryan L, Chitra S, Noble R, McGovern PC. Safety and efficacy of omadacycline for treatment of community-acquired bacterial pneumonia and acute bacterial skin and skin structure infections in patients with mild-to-moderate renal impairment. Int J Antimicrob Agents. 2021 Feb;57(2):106263. doi: 10.1016/j.ijantimicag.2020.106263. Epub 2020 Dec 14. PMID 33326848
- [Derived] O'Riordan W, Cardenas C, Shin E, Sirbu A, Garrity-Ryan L, Das AF, Eckburg PB, Manley A, Steenbergen JN, Tzanis E, McGovern PC, Loh E; OASIS-2 Investigators. Once-daily oral omadacycline versus twice-daily oral linezolid for acute bacterial skin and skin structure infections (OASIS-2): a phase 3, double-blind, multicentre, randomised, controlled, non-inferiority trial. Lancet Infect Dis. 2019 Oct;19(10):1080-1090. doi: 10.1016/S1473-3099(19)30275-0. Epub 2019 Aug 29. PMID 31474458
- [Derived] Abrahamian FM, Sakoulas G, Tzanis E, Manley A, Steenbergen J, Das AF, Eckburg PB, McGovern PC. Omadacycline for Acute Bacterial Skin and Skin Structure Infections. Clin Infect Dis. 2019 Aug 1;69(Suppl 1):S23-S32. doi: 10.1093/cid/ciz396. PMID 31367742

RESULTS

PARTICIPANT FLOW:
Groups:
- Omadacycline: Participants received omadacycline 450 milligrams (mg) orally every 24 hours (q24h) for 2 doses, followed by 300 mg orally q24h. The total treatment duration was 7 to 14 days. Participants received active omadacycline tablets and over-encapsulated linezolid placebo tablets.
- Linezolid: Participants received linezolid 600 mg orally every 12 hours (q12h). The total treatment duration was 7 to 14 days. Participants received omadacycline placebo tablets and over-encapsulated active linezolid tablets.
Period: Overall Study
Arm/Group | Omadacycline | Linezolid
Started | 368 | 367
Completed | 314 | 310
Not Completed | 54 | 57
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 37 | 38
Not completed — Withdrawal by Subject | 11 | 12
Not completed — Physician Decision | 0 | 1
Not completed — Missed EOT/PTE Visit | 5 | 6

BASELINE CHARACTERISTICS:
Population: Safety Population: all randomized participants who received test article
Groups:
- Total: Total of all reporting groups
Arm/Group | Omadacycline | Linezolid | Total
Number analyzed (Participants) | 368 | 367 | 735
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (12.72) | 44.5 (13.11) | 43.7 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 147 | 273
  Male | 242 | 220 | 462
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 3 | 10
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 22 | 13 | 35
  White | 327 | 341 | 668
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Early Clinical Response
Description: Early clinical response is defined as clinical success, which is categorized as survival with at least a 20% reduction of acute bacterial skin and skin structure infection (ABSSSI) primary lesion size compared to Screening measurements, without receiving any rescue antibacterial therapy. An indeterminate classification is used for a response that could not be adequately inferred because the participant was not assessed because they withdrew consent, were lost to follow-up, or other specified reason.
Time Frame: Screening; 48 to 72 hours after the first dose of test article
Population: Modified Intent-to-Treat (mITT) Population: all randomized participants without a baseline sole Gram-negative ABSSSI pathogen
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 360 | 360
Participants
  Clinical success | 315 | 297
  Clinical failure | 26 | 32
  Indeterminate | 19 | 31
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = 5.0, 95% CI 2-sided [-0.2 to 10.3] — The 95% confidence interval was constructed based on the Miettinen and Nurminen method without stratification. Treatment difference for a response of clinical success was calculated as omadacycline minus linezolid

2. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Clinical Response in the mITT Population at the Post Therapy Evaluation (PTE) Visit
Description: At the PTE Visit the investigator indicated one of the following outcomes relating to the primary infection under study: Clinical Success: participant was alive; infection was sufficiently resolved such that further antibacterial therapy was not needed. Participants may have had some residual changes related to infection requiring ancillary treatment. Clinical Failure was defined as meeting any of the following criteria: infection required additional treatment with alternative antibacterial therapy; participant received antibacterial therapy between the End-of-Treatment (EOT) Visit and the PTE Visit that may have been effective for the infection under study for a different infection from the one under study; unplanned major surgical intervention for the infection under study between the EOT and PTE Visits; participant died before evaluation; other specified reason. Indeterminate The clinical response to test article could not be adequately inferred.
Time Frame: Screening; 7 to 14 days after the last day of therapy
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 360 | 360
Participants
  Clinical success | 303 | 291
  Clinical failure | 12 | 21
  Indeterminate | 45 | 48
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = 3.3, 95% CI 2-sided [-2.2 to 8.9] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Clinical Response in the Clinically Evaluable-Post Therapy Evaluation (CE-PTE) Population
Description: At the PTE Visit the investigator indicated one of the following outcomes relating to the primary infection under study: Clinical Success: participant was alive; infection was sufficiently resolved such that further antibacterial therapy was not needed. Participants may have had some residual changes related to infection requiring ancillary treatment. Clinical Failure was defined as meeting any of the following criteria: infection required additional treatment with alternative antibacterial therapy; participant received antibacterial therapy between the EOT Visit and the PTE Visit that may have been effective for the infection under study for a different infection from the one under study; unplanned major surgical intervention for the infection under study between the EOT and PTE Visits; participant died before evaluation; other specified reason.
Time Frame: Screening; 7 to 14 days after the last day of therapy
Population: CE-PTE Population: all participants in the mITT Population meeting additional pre-defined criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 284 | 292
Participants
  Clinical success | 278 | 279
  Clinical failure | 6 | 13
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = 2.3, 95% CI 2-sided [-0.6 to 5.6] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the signing of Informed Consent Form to the time of the Final Follow-up assessment (up to 30 to 37 days after the first dose of test article).
Description: Adverse events are reported for members of the Safety Population, comprised of all randomized participants who received test article (either active or placebo). Treatment-emergent adverse events, defined as events occurring after the first dose of active test article, are reported.
Arm/Group | Omadacycline | Linezolid
All-Cause Mortality (participants affected / at risk) | 0/368 | 1/367
Serious Adverse Events (participants affected / at risk) | 5/368 | 5/367
Other Adverse Events (participants affected / at risk) | 166/368 | 83/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=368) | Linezolid (N=367)
Drug Withdrawal Syndrome (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=368) | Linezolid (N=367)
Nausea (Gastrointestinal disorders) | 111 | 28
Vomiting (Gastrointestinal disorders) | 62 | 11
Diarrhea (Gastrointestinal disorders) | 15 | 10
Abdominal pain upper (Gastrointestinal disorders) | 10 | 4
Wound infection (Infections and infestations) | 21 | 16
Cellulitis (Infections and infestations) | 12 | 8
Subcutaneous abscess (Infections and infestations) | 5 | 8
Alanine aminotransferase increased (Investigations) | 19 | 11
Aspartate aminotransferase increased (Investigations) | 17 | 12
Headache (Nervous system disorders) | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the Principal Investigator is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can request changes to the communication and require the removal of confidential information.

DOCUMENTS (2):
  • Study Protocol (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT02877927/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT02877927/SAP_001.pdf